CLINICAL TRIAL: NCT05397015
Title: Metabotyping in the Postmenopausal Stage: Cross-Sectional Observational Study
Brief Title: Metabotyping in the Postmenopausal Stage
Acronym: SHE-HEALTH
Status: Completed | Type: Observational
Sponsor: Fundació Eurecat (Other)
Responsible Party: Sponsor
Other Study IDs: SHE-HEALTH
Record Dates: First submitted 2022-04-01; First posted 2022-05-31 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Menopause; Postmenopausal Disorder; Postmenopausal Symptoms
Keywords: Metabolomics; Transcriptomics; Metagenomics; Personalized Nutrition; Metabotypes; Enterotypes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of blood, faeces, urine, hair and hair follicles will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postmenopausal women: A cohort of 200 postmenopausal women
  Interventions: Other: No intervention will be done

INTERVENTIONS:
Other: No intervention will be done — No intervention will be done

SUMMARY:
Menopause is defined as the absence of menstrual periods for twelve consecutive months. Although the onset may vary, natural menopause occurs between the ages of 45 and 55 and is considered a stage in the aging process for women. Menopause is a stage strongly conditioned by hormonal modulations with effects on the cardiovascular system associated with abdominal obesity, insulin resistance, decreased energy expenditure, endothelial dysfunction, hypertension, and dyslipidemia. Furthermore, an increase in the production of proinflammatory cytokines involved in numerous pathologies such as osteoporosis has been observed.

The results of several studies suggest that intestinal microbiota (IM) profile may be related to menopause condition by several means, although the data are stil inconclusive.

Estrogen reduction leads to a progressive loss of bone density, a reduction in the bone formation/resorption balance and an increased risk of bone fractures among postmenopausal women. Recently, the alternative to estrogen therapies to reduce the risk of fractures are nutritional strategies fundamentally based on the use of probiotics, whose effect are associated with beneficial modulations of IM.

SHE-HEALTH is a study in which, in a cohort of postmenopausal women, metabolomics, transcriptomics and metagenomics will be combined with the analysis of usual anthropometric and clinical biomarkers and also with genetic and epigenetic analyses to identify population groups (clusters). This study will allow establishing solid scientific bases to define, in future projects, effective nutritional strategies based on group nutrition in postmenopausal women.

The main objective of the present study is to obtain clusters of postmenopausal women, identifying metabotypes (similar metabolic profiles) and enterotypes (similar IM profiles), and combining complementary variables such as classical anthropometric, biochemical and clinical biomarkers.

The secondary objectives of the study are to characterize: 1) The genetic profile of the study cohort; 2) The epigenetic profile of the study cohort; 3) The gene expression profile of the study cohort.

DETAILED DESCRIPTION:
Cross-sectional observational study in which samples of blood, faeces, urine, hair and hair follicles will be collected to characterize the metabolic profile, intestinal microbiota (IM), gene expression profile, genetic and epigenetic profile of postmenopausal women. Data on lifestyle habits, anthropometric measurements and nutritional and hormonal status will also be collected.

The study will be conducted in a cohort of 200 postmenopausal women.

Each volunteer will make 2 visits:

* A pre-selection visit (to check inclusion/exclusion criteria) (V0) and, if the inclusion criteria are met,
* A study visit (V1) in which samples will be collected from faeces, urine, blood, hair and hair follicles.

In V1, the participants must present themselves fasting for 8 hours to obtain blood and urine collected during the last 24 hours. In addition, during the visit the sample of hair and hair follicles will be collected. Participants are given a basic guide of healthy eating and lifestyle recommendations suitable for postmenopausal stage.

ELIGIBILITY:
Inclusion Criteria:

* Women between 40 and 63 years old with amenorrhea for a period of time equal or greater than 12 months.
* Without hormone replacement therapy.
* Sign the informed consent.

Exclusion Criteria:

* Women diagnosed with diabetes (or serum glucose ≥ 126 mg/dL) or other chronic pathologies (coronary, cardiovascular, celiac disease, Crohn's disease and chronic kidney diseases (or serum creatinine ≥ 1.5 mg/dL).
* Women taking medications prescribed for hypertension and dyslipidemia. Women who have consumed during the week prior to start to start of the study anti-inflammatory drugs.
* women with chronic gastrointestinal problems.
* Women with a body mass index (in kg/m2) <18 or ≥35.
* Women who are participating in another clinical trial or following a prescribed diet for any reason, including weigh loss, during the last month.
* Women who consume more than 14 alcoholic beverages per week.
* Women current smokers.

Ages: 40 Years to 63 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The cohort of the study will be selected from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Metabolomics in serum | At day 1
  Non-targeted metabolomics of serum samples measured using proton nuclear magnetic resonance. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Metabolomics in erythrocytes | At day 1
  Non-targeted metabolomics of erythrocytes samples measured using proton nuclear magnetic resonance. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Metabolomics in urine | At day 1
  Non-targeted metabolomics of urine samples measured using proton nuclear magnetic resonance. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Metagenomics in faeces | At day 1
  Faecal intestinal microbiota analysis will be done by 16sRNA sequencing. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum hsCRP levels | At day 1
  Serum hsCRP levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum IL-6 levels | At day 1
  Serum IL-6 levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum TNFalpha levels | At day 1
  Serum TNFalpha levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum BALP levels | At day 1
  Serum BALP levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum osteocalcin levels | At day 1
  Serum osteocalcin levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum TRAP5b levels | At day 1
  Serum TRAP5b levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum CTX-I levels | At day 1
  Serum CTX-I levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum PINP levels | At day 1
  Serum PINP levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum FSH levels | At day 1
  Serum FSH levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum 17beta E2 levels | At day 1
  Serum 17beta E2 levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum inhibin B levels | At day 1
  Serum inhibin B levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum testosterone levels | At day 1
  Serum testosterone levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum AMH levels | At day 1
  Serum AMH levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum SHBG levels | At day 1
  Serum SHBG levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum triglycerides levels | At day 1
  Serum triglycerides levels will be measured by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum total cholesterol levels | At day 1
  Serum total cholesterol levels will be measured by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum LDL-cholesterol levels | At day 1
  Serum LDL-cholesterol levels will be measured by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum HDL-cholesterol levels | At day 1
  Serum HDL-cholesterol levels will be measured by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum glucose levels | At day 1
  Serum glucose levels will be measured by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum insulin levels | At day 1
  Serum insulin levels will be measured by Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Homeostatic Model Assessment from Insulin Resistance index (HOMA-IR) | At day 1
  HOMA-IR will be calculated using serum glucose and insulin levels. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum ALT levels | At day 1
  Serum ALT levels will be measured by Cobas Mira Plus autoanalyzer (RocheDiagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum AST levels | At day 1
  Serum AST levels will be measured by Cobas Mira Plus autoanalyzer (RocheDiagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum creatinine levels | At day 1
  Serum creatinine levels will be measured by Cobas Mira Plus autoanalyzer (RocheDiagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum uric acid levels | At day 1
  Serum uric acid levels will be measured by Cobas Mira Plus autoanalyzer (RocheDiagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Serum urea levels | At day 1
  Serum urea levels will be measured by Cobas Mira Plus autoanalyzer (RocheDiagnostics Systems, Madrid, Spain). Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Urine 8-OHdG levels | At day 1
  Urine 8-OHdG levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Urine F2-isoprostanes levels | At day 1
  Urine F2-isoprostanes levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.
Urine NTX levels | At day 1
  Urine NTX levels will be measured by human ELISA kits. Data will be analysed together with the other primary outcomes for cluster identification. Data will be scaled using unit variance scaling. Principal components analysis, Partial Least-Squares Discriminant Analysis and hierarchical clustering will be used to identify clusters and to detect differences among metabotypes. The quality of the model will be judged by the goodness-of-fit parameter, the predictive ability parameter and cross-validation test.

SECONDARY OUTCOMES:
Body weight | At day 1
  Body weight measured by TANITA SC 330 S portable scale (Peroxfarma, Barcelona, Spain) .
Height | At day 1
  Height measured by TANITA Leicester Portable (Tanita Corp., Barcelona, Spain)
Body mass index | At day 1
  Weight and height will be combined to report body mass index in kg/m^2
Waist circumference | At day 1
  Waist circumference will be measured using a 150 cm anthropometric steel measuring tape
Blood pressure (in mmHg) | At day 1
  Systolic and diastolic pressure will be measured twice after 2-5 minutes of patient respite, seated, with one minute interval in between, using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Waist circumference to height ratio | At day 1
  Waist circumference and height will be combined to report waist circumference to height ratio.
Body composition | At day 1
  Body fat mass and body lean mass will be measured using TANITA SC 330 S Body Composition Analyzer (Peroxfarma, Barcelona, Spain)
Dietary intake | At day 1
  Dietary intake will be measured using 3-day dietary record.
Transcriptomics analysis in hair follicles. | At day 1
  Transcriptomics analysis in hair follicles samples will be done by RNA-seq.
Transcriptomics analysis in total blood. | At day 1
  Transcriptomic analysis will be performed with blood samples collected in PAXgene tubes by microarray technology (Agilent Technologies). This analysis will be carried out with a sub-cohort of post-menopausal women from each of the different clusters obtained with a total of 64 samples.
MicroRNAs analysis in total blood. | At day 1
  MicroRNAs will be analyzed in blood samples collected in PAX gene tubes using RNA-seq technology. This analysis will be carried out with a sub-cohort of post-menopausal women from each of the different clusters obtained with a total of 64 samples.
DNA methylation analysis in total blood. | At day 1
  DNA methylation analysis will be performed with blood samples collected in PAXgene tubes by bisulfite conversion of the DNA combined with targeted amplification of regions of interest, library construction and next-generation sequencing. This analysis will be carried out with a sub-cohort of post-menopausal women from each of the different clusters obtained with a total of 64 samples.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — Eurecat-Reus
Locations (1):
- Eurecat, Reus, Spain

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org